CLINICAL TRIAL: NCT05778032
Title: Biological Age Assessment in Adults With Prader-Willi Syndrome Undergoing an Integrated Multidisciplinary Metabolic Rehabilitation Program
Brief Title: Biological Age Assessment in Adults With Prader-Willi Syndrome (ETABIOLPWS)
Acronym: ETABIOLPWS
Status: Active, not recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C213
Record Dates: First submitted 2023-02-26; First posted 2023-03-21 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Obesity; Biological age; Metabolic rehabilitation
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples taken will be used for DNA extraction. DNA methylation will be performed by treatment with sodium bisulphite and PCR-Pyrosequencing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multidisciplinary metabolic rehabilitation program — Multidisciplinary metabolic rehabilitation program with a duration of 3 weeks

SUMMARY:
The primary objective of the study is to compare, in a cohort of obese subjects with PWS hospitalized at the Division of Auxology, Istituto Auxologico Italiano, Piancavallo (VB), Italy, the age acceleration calculated at study entry (T0) with the age acceleration measured at the end of a 3-week multidisciplinary metabolic rehabilitation program (T1).

Secondary objectives are to correlate the biological age with the anthropometric characteristics (with particular reference to the body composition), the glycometabolic picture, the main parameters and cardiovascular risk factors, the therapy (previous and concomitant) with rhGH and the cognitive function (mainly, the IQ).

DETAILED DESCRIPTION:
Methods Thirty adults affected by clinically diagnosed and genetically confirmed PWS are recruited, regardless of the treatment (previous or concomitant) with rhGH (F/M = 15/15; age: ≥ 18 years; BMI > 35 kg/m2), hospitalized for a period of integrated multidisciplinary metabolic rehabilitation at the Division of Auxology, Istituto Auxologico Italiano, Piancavallo (VB), Italy.

After verifying the inclusion criteria, clinical and anthropometric data will be collected, including the evaluation of body composition with bioimpedance analysis. Cognitive function will be assessed with a psychometric scale (Wechsler Adult Intelligence Scale).

Blood samples will be taken from each patient upon admission to the hospital (T0) and after 3 weeks of rehabilitation hospitalization (at the same time to reduce circadian variability) for the determination of the basal glycometabolic profile (glucose, insulin, HOMA-IR, glycated Hb , triglycerides, total cholesterol, LDL, HDL, and hsPCR), as well as circulating levels of leptin, IL-6, and TNF-α.

The samples taken will be used for DNA extraction. DNA methylation will be performed by treatment with sodium bisulphite and PCR-Pyrosequencing.

Biological age measurement Biological (epigenetic) age will be measured using the two algorithms of Zbiec-Piekarska (9) and Daunay (10), based on the level of DNA methylation in specific gene loci. To have an estimate of the epigenetic (biological) age that is independent of the chronological age, we will use a measure defined as age acceleration, from which, with statistical inference, we will calculate the age acceleration. To calculate it, a linear regression model with the chronological age as the independent variable and the epigenetic age as the dependent variable will be applied; the difference between the observed value and the one predicted by the model will constitute the age acceleration due to epigenetic effects. In the event that the epigenetic age is greater than the chronological age, the age acceleration will have a positive value expressed in years, negative if vice versa.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with PWS, clinically diagnosed and genetically confirmed, regardless of rhGH treatment (previous or concomitant)
* age: ≥ 18 years
* BMI > 35 kg/m2
* hospitalization for integrated multidisciplinary metabolic rehabilitation program

Exclusion Criteria:

* age < 18 years
* BMI < 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with Prader-Willi syndrome with BMI > 35 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DNA methylation | Baseline and at the end of the rehabilitation program (21 days)
  Change in level of DNA methylation

SECONDARY OUTCOMES:
Glycometabolic profile: glucose | Baseline and at the end of the rehabilitation program (21 days)
  Change in glycometabolic profile - glucose levels
Glycometabolic profile: insulin | Baseline and at the end of the rehabilitation program (21 days)
  Change in glycometabolic profile - insulin levels
Body fat mass | Baseline and at the end of the rehabilitation program (21 days)
  Change in body fat mass - bioimpedance analysis
Body fat free mass | Baseline and at the end of the rehabilitation program (21 days)
  Change in body fat free mass - bioimpedance analysis
Body weight | Baseline and at the end of the rehabilitation program (21 days)
  Change in body weight
Body mass index | Baseline and at the end of the rehabilitation program (21 days)
  Change in body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy